CLINICAL TRIAL: NCT02898337
Title: Methadone-Induced QT Interval Prolongation in a Narcotic Treatment Center: Identifying Patients at Risk and Simplifying ECG Monitoring
Brief Title: Methadone-Induced QT Interval Prolongation in a Narcotic Treatment Center
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, James E. Tisdale, Adjunct Professor, Indiana University
Other Study IDs: 1608001774
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: QT Interval Prolongation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples for determination of cytochrome P-450 2B6 genotype
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Methadone-induced QTc interval prolongation
  Interventions: Device: AliveCor handheld mobile ECG
- Methadone-treated patients, no QT interval prolongation
  Interventions: Device: AliveCor handheld mobile ECG

INTERVENTIONS:
Device: AliveCor handheld mobile ECG — Specific Aim 1: independent risk factors for methadone-associated QTc interval prolongation will be determined through retrospective analysis of electronic medical records of methadone-treated patients in a narcotic treatment center. Patients will be asked to come to the Narcotic Treatment Center for one 12-lead ECG
  Specific Aim 2: QTc intervals from ECGs generated by the AliveCor® heart monitor will be compared prospectively to simultaneous twelve lead ECGs for validation purposes in the methadone-treated patients in a narcotic treatment center.

SUMMARY:
Torsades de pointes (TdP) is a polymorphic ventricular tachycardia associated with prolongation of the heart rate-corrected QT (QTc) interval on the electrocardiogram (ECG). TdP can result in catastrophic outcomes, including sudden cardiac death. QTc interval prolongation is a well-known adverse event associated with methadone use. While some risk factors for methadone-associated QTc interval prolongation and TdP have been identified, the contribution of interacting drugs and concomitant administration of other QTc interval-prolonging agents to overall risk has not been determined. The effect of ECG screening and monitoring on clinical outcomes in patients taking methadone has not been evaluated, and clinical opinion regarding routine ECG and risk factor monitoring varies. Twelve lead ECGs are costly and time-intensive for clinic staff. ECG screening in selected patients based on presence of QTc interval risk factors, rather than broadly in all patients taking methadone, would facilitate more targeted, strategic QTc interval monitoring. The FDA-approved AliveCor® handheld smart phone/tablet device records a single lead ECG (iECG) within 30 seconds. Use of this device may facilitate simpler, more rapid and less costly ECG monitoring in patients receiving care in narcotic treatment centers.

Our long-term goals are to determine mechanisms by which drugs cause arrhythmias, to identify patients at greatest risk of drug-induced arrhythmias, and to determine safe and effective methods for prevention and management of drug-induced arrhythmias.

Specific Aim 1: Identify independent risk factors for methadone-induced QTc interval prolongation in patients undergoing care in a narcotic treatment center.

Research Design: This will be a retrospective/prospective analysis of ECGs and health information from patients receiving methadone therapy in the Eskenazi Health Midtown Narcotic Treatment Center in Indianapolis, IN. Currently, at the Midtown Narcotic Treatment Center, baseline 12-lead ECGs are recorded for all patients prior to initiation of methadone therapy; follow-up ECGs are obtained approximately 2 weeks after methadone initiation only in patients with a baseline prolonged QTc interval. At the start of the study, methadone-treated patients who have not had follow-up ECGs on methadone therapy will be identified and contacted prospectively. Those consenting to participation will undergo a follow-up 12-lead ECG to determine QTc interval during methadone maintenance therapy. For all patients, retrospective analysis of the electronic medical record will be performed to document sex, pregnancy status, age, family history, current and past medical history, and concomitant use of prescribed, over the counter, and illicit drug use with the aim to identify all potential risks. QTc interval prolongation will be defined as QTc interval ≥ 500 ms or an increase in QTc interval of ≥ 60 ms compared with the baseline QTc interval. Electronic health information variables will be compared in patients who develop methadone-associated QTc interval prolongation versus those who do not using univariate analysis. Patients with prolonged QTc interval at baseline will be excluded from the study.

Specific Aim 2: Validate the handheld AliveCor® smart phone/tablet iECG device as a simple, rapid method of monitoring QTc intervals in methadone-treated patients in a narcotic treatment center.

Research Design: A separate cohort of patients will be utilized to validate the AliveCor® device for use in measuring QTc intervals in patients initiated and maintained on methadone in a narcotic treatment center. Twelve lead ECGs and simultaneous single lead ECGs using the AliveCor® device will be recorded for all newly enrolled patients at baseline and again after six weeks of methadone therapy. The QTc identified by the 12-lead ECG will be compared to the single lead ECG for all baseline and follow-up recordings to validate the use of the AliveCor® device for potential use in narcotic treatment centers to reduce cost and save time. Comparison of QTc intervals between the 12-lead and single lead measurements will be performed using the Bland-Altman method for analysis of measurement agreement. The mean and 95% confidence interval of the difference in QTc interval between the two methods will be calculated.

This will be a pilot study to justify a larger extramural study to develop and validate a risk score for methadone-induced QTc interval prolongation and to use the handheld ECG device for QTc interval monitoring in patients identified as high-risk using this risk score. Our rationale is that identification of risk factors for methadone-induced QTc interval prolongation and quantification of degree of risk conferred by each risk factor will ultimately reduce the incidence and risk of QTc interval prolongation through targeted ECG monitoring of patients at highest risk and modulation of modifiable risk factors.

DETAILED DESCRIPTION:
Specific Aims:

Torsades de pointes (TdP) is a polymorphic ventricular tachycardia associated with prolongation of the heart rate-corrected QT (QTc) interval on the electrocardiogram (ECG). TdP can result in catastrophic outcomes, including sudden cardiac death. QTc interval prolongation is a well-known adverse event associated with methadone use. While some risk factors for methadone-associated QTc interval prolongation and TdP have been identified, the contribution of interacting drugs and concomitant administration of other QTc interval-prolonging agents to overall risk has not been determined. The effect of ECG screening and monitoring on clinical outcomes in patients taking methadone has not been evaluated, and clinical opinion regarding routine ECG and risk factor monitoring varies. The Methadone Safety Guidelines, detailed in the Research Strategy, do not provide clear recommendations for baseline and follow-up ECGs. Twelve lead ECGs are costly and time-intensive for clinic staff. ECG screening in selected patients based on presence of QTc interval risk factors, rather than broadly in all patients taking methadone, would facilitate more targeted, strategic QTc interval monitoring. The FDA-approved AliveCor® handheld smartphone/tablet device records a single lead ECG (iECG) within 30 seconds. Use of this device may facilitate simpler, more rapid and less costly ECG monitoring in patients receiving care in narcotic treatment centers. Identification of QTc interval prolongation risk factors in patients receiving methadone in a narcotic treatment center will enable early identification of patients at risk for QTc interval prolongation, so that modifiable risk factors may be addressed and ECG monitoring intensified to reduce the odds of patients progressing to develop methadone-associated QTc interval prolongation with the attendant risk of TdP.

Our long-term goals are to determine mechanisms by which drugs cause arrhythmias, to identify patients at greatest risk of drug-induced arrhythmias, and to determine safe and effective methods for prevention and management of drug-induced arrhythmias. The short-term goal in this application is to identify independent risk factors for methadone-induced QTc interval prolongation in patients undergoing care in a narcotic treatment center and to validate the use of the handheld AliveCor® iECG as a method for screening and monitoring for methadone-induced QTc interval prolongation in this patient population. Our central hypothesis is that identification and management of risk factors and use of the AliveCor® iECG to screen and monitor patients initiated and maintained on methadone in a narcotic treatment center will reduce the risk of QTc interval prolongation. In this pilot study, the investigators propose the following specific aims:

Specific Aim 1: Identify independent risk factors for methadone-induced QTc interval prolongation in patients undergoing care in a narcotic treatment center.

Hypothesis: Risk factors for methadone-associated QTc interval prolongation include female sex, older age, methadone dose, receiving at least one additional QTc interval prolonging medication, concomitant therapy with diuretics, and concomitant therapy with drugs that are cytochrome P-450 2B6 inhibitors, including clopidogrel, ticlopidine and voriconazole. To test this hypothesis, independent risk factors for methadone-associated QTc interval prolongation will be determined through retrospective analysis of electronic medical records of methadone-treated patients in a narcotic treatment center.

Specific Aim 2: Validate the handheld AliveCor® smartphone/tablet iECG device as a simple, rapid method of monitoring QTc intervals in methadone-treated patients in a narcotic treatment center.

Hypothesis: The AliveCor® handheld smartphone/tablet iECG device is a valid method of measuring QTc intervals in methadone-treated patients. To test this hypothesis, QTc intervals from ECGs generated by the AliveCor® heart monitor will be compared prospectively to simultaneous twelve lead ECGs for validation purposes in the methadone-treated patients in a narcotic treatment center.

The proposed work will be a pilot study to justify a larger extramural study to develop and validate a risk score for methadone-induced QTc interval prolongation and to use the handheld ECG device for QTc interval monitoring in patients identified as high-risk using this risk score. Our rationale is that identification of risk factors for methadone-induced QTc interval prolongation and quantification of degree of risk conferred by each risk factor will ultimately reduce the incidence and risk of QTc interval prolongation through targeted ECG monitoring of patients at highest risk and modulation of modifiable risk factors. Our expected outcome is that independent risk factors for methadone-induced QTc interval prolongation will be identified, and that the AliveCor® handheld iECG device will perform as well as 12-lead ECGs for assessing QTc intervals in methadone-treated patients.

Research Plan:

Specific Aim 1: Identify independent risk factors for methadone-induced QTc interval prolongation in patients undergoing care in a narcotic treatment center.

This will be a retrospective/prospective analysis of ECGs and health information from patients receiving methadone therapy in the Eskenazi Health Midtown Narcotic Treatment Center in Indianapolis, IN. This center is one of Eskenazi Health Midtown's outpatient specialty substance abuse centers which employs a treatment team consisting of an addiction psychiatrist, nurses, licensed addiction counselors, and case managers. The center serves over 1,000 patients each year, and there are between 250 and 300 patients receiving methadone treatment in the center at any given time. Currently, at the Midtown Narcotic Treatment Center, baseline 12-lead ECGs are recorded for all patients prior to initiation of methadone therapy; follow-up ECGs are obtained approximately 2 weeks after methadone initiation only in patients with a baseline prolonged QTc interval. Patients with prolonged QTc interval at baseline will be excluded from the study.

At the start of the study, methadone-treated patients who have not had follow-up ECGs on methadone therapy will be identified and contacted prospectively. Those consenting to participation will undergo a follow-up 12-lead ECG to determine QTc interval during methadone maintenance therapy.

For all patients, retrospective analysis of electronic medical record will be performed to document sex, pregnancy status, age, family history, current and past medical history, and concomitant use of prescribed, over the counter, and illicit drug use with the aim to identify all potential risks. The Credible Meds database will be referenced to identify all QTc interval-prolonging medications with a known or possible risk of TdP.60 There are currently 165 medications identified by Credible Meds to have a known or possible risk, and this list will be accessed again at the start of study in the case any new medications have been added.

QT intervals will be measured from leads II, V1, and V5 by one investigator (ET-L) who will be blinded to baseline vs on-treatment status. QT intervals will be measured using the MUSE automated system (GE Healthcare Bio-Sciences, Pittsburgh, PA) using electronic calipers. QT and RR intervals will be averaged over ≥ 5 consecutive beats and the average of three QT intervals at each time point for each lead will be determined. Only clearly discernible QT intervals will be measured. QT intervals will be corrected for heart rate using Bazett's formula:61

While Bazett's formula has some limitations, the investigators will use this correction in this study because it is standard of practice for QTc interval monitoring for patient care purposes, and there are no accepted definitions of QTc interval prolongation using other heart rate correction factors. QTc interval prolongation will be defined as QTc interval ≥ 500 ms or an increase in QTc interval of ≥ 60 ms compared with the admitting value at any time during hospitalization.62,63

Electronic health information variables will be compared in patients who develop methadone-associated QTc interval prolongation versus those who do not using univariate analysis. Unpaired Student's t-test will be used to compare continuous variables, assuming equal or unequal variances between the groups, and Chi-Square or Fisher's Exact test, as appropriate, will be used for categorical variables. Comparisons for non-normally distributed continuous parameters will be performed using the non-parametric Wilcoxon Rank Sum test. In order to determine independent predictors of QTc interval prolongation, univariate variables with a p value ≤ 0.10 will be incorporated into a bivariate logistic regression model in a forward stepwise fashion in descending order of those most strongly associated with QTc interval prolongation based on univariate p value. Significant continuous variables will be dichotomized based on the results of the univariate analysis. Dichotomized variables will be compared using the Chi square or Fisher's Exact test as appropriate. Odds ratios (OR) with 95% confidence intervals (CI) will be determined for each variable. Statistical analyses will be performed using SPSS 24.0 (SPSS, Inc., Chicago, IL, USA).

Specific Aim 2: Validate the handheld AliveCor® smartphone/tablet iECG device as a simple rapid method of monitoring QTc intervals in methadone-treated patients in a narcotic treatment center.

The second specific aim will utilize a separate cohort of patients to validate the AliveCor® device for use in measuring QTc intervals in patients initiated and maintained on methadone in a narcotic treatment center. Approximately 20 to 30 new patients are enrolled each month in the Eskenazi Health Midtown Narcotics Treatment Center. Data collection will be completed over the course of two months with the aim to enroll 40 to 60 patients for this aim. Twelve lead ECGs (Marquette Mac 5500, GE Healthcare Bio-Sciences, Pittsburgh, PA) and simultaneous single lead ECGs using the AliveCor® device will be recorded for all newly enrolled patients at baseline and again after six weeks of methadone therapy. The QTc identified by the twelve lead ECG will be compared to the single lead ECG for all baseline and follow-up recordings to validate the use of the AliveCor® device for potential use in narcotic treatment centers to reduce cost and save time. The single lead ECG will be uploaded to a computer and measured manually by study researchers using ECG calipers. QT intervals will be measured and corrected as described previously.

A total of 80 to 120 QTc intervals, depending on the number of patients enrolled, will be compared. Comparison of QT intervals between the twelve lead and single lead measurements will be performed using the Bland-Altman method for analysis of measurement agreement. The mean and 95% confidence interval of the difference in QT interval between the two methods will be calculated. Logistic regression analysis will be utilized to identify independent predictors of perfect agreement between both measurements, where perfect agreement is defined as agreement within 20 ms between the two measurements. Odds ratios and 95% confidence intervals of each independent predictor will be calculated. Using the twelve lead ECG as the gold standard, the sensitivity and specificity of the single lead ECG will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the Eskenazi Health Midtown Narcotic Treatment Center between August 1, 2014 - December 31, 2016
* 18 years and older

Exclusion Criteria:

* Documented history by prescriber or baseline prolonged QTc interval
* Patients with insufficient information in the electronic health record
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing methadone treatment for addiction in a narcotic treatment center
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
QTc interval prolongation | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Eskenazi Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Titus-Lay EN, Jaynes HA, Tomaselli Muensterman E, Ott CA, Walroth TA, Williams G, Moe PR, Wilbrandt M, Tisdale JE. Accuracy of a single-lead mobile smartphone electrocardiogram for QT interval measurement in patients undergoing maintenance methadone therapy. Pharmacotherapy. 2021 Jun;41(6):494-500. doi: 10.1002/phar.2521. Epub 2021 Apr 19. PMID 33772822
- [Derived] Titus-Lay EN, Jaynes HA, Tomaselli Muensterman E, Walroth TA, Ott CA, Desta Z, Williams G, Moe PR, Wilbrandt M, Tisdale JE. Methadone-associated QT interval prolongation in patients undergoing maintenance therapy in an urban opioid treatment program. Pharmacotherapy. 2021 Mar;41(3):238-246. doi: 10.1002/phar.2498. Epub 2021 Feb 2. PMID 33345336